CLINICAL TRIAL: NCT04236050
Title: Comparison of the Effect of Continuous Infusion and Bolus Doses of Rocuronium During Anesthesia for Lumbal Discectomy on Muscle Strength and Quality of Patient Recovery
Brief Title: Continuous Infusion and Bolus Doses of Rocuronium During Lumbal Discectomy, Muscle Strength and Patient Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Martina Miklic Bublic, MD, PhD, Principal Investigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 021
Record Dates: First submitted 2020-01-09; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Rocuronium; Lumbar Discectomy; Recovery
Keywords: rocuronium; Qor-40; lumbar discectomy; muscle strength
MeSH Terms: interventions — Rocuronium; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rocuronium is administered via continuous infusion (Experimental): 40 patients. General anesthesia is maintained with propofol and remifentanil, with standard anesthetic monitoring, bispectral index (BIS) and train-of-four(TOF). In experimental group, rocuronium was administered via continuous infusion so that theTOF ratio was 5%. Hand-grip muscle strength was measured with a dynamometer on three occasions: before general anesthesia, in the early post-anesthesia period in the operating room, and 24 hours after anesthesia.
  The quality of patient recovery was assessed with a Qor-40 questionnaire before anesthesia, 24 hours after anesthesia, and 30 days after anesthesia and surgery
  Interventions: Drug: Rocuronium
- rocuronium is administered in bolus doses (Active Comparator): 40 patients. General anesthesia was maintained with propofol and remifentanil, with standard anesthetic monitoring, BIS and TOF. In this group, rocuronium was administered in separate bolus doses with the TOF ratio of 5%.
  Hand-grip muscle strength was measured with a dynamometer on three occasions: before general anesthesia, in the early post-anesthesia period in the operating room, and 24 hours after anesthesia.
  The quality of patient recovery was assessed with a Qor-40 questionnaire before anesthesia, 24 hours after anesthesia, and 30 days after anesthesia and surgery
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Rocuronium administered in continuous infusion or multiple bolus doses
  Other Names: general anesthesia

SUMMARY:
The continuous infusion of rocuronium during general anesthesia for a lumbar discectomy enables better muscle strength recovery, and a better quality of patient recovery as measured by questionnaire.

DETAILED DESCRIPTION:
Rocuronium is a non-depolarising neuromuscular blocking agent that can be administered in bolus doses or via continuous infusion during general anesthesia. Due to the specificity of the knee-chest position in a lumbar discectomy, many complications during anesthesia and surgery are possible. Therefore an effective and balanced intraoperative neuromuscular block is needed.

Studies so far have not included a comparison on muscle strength and quality of patient recovery of the effect of continuous infusion and bolus doses of rocuronium during anesthesia for lumbar discectomy.

The hypothesis of this research was that the continuous infusion of rocuronium during general anesthesia for a lumbar discectomy enables better muscle strength recovery, and a better quality of patient recovery as measured by questionnaire.

The aim was to compare the influence of the continuous infusion and bolus doses of rocuronium on patient recovery. Therefore the investigators assessed how continuous infusion and bolus doses of rocuronium affect the recovery of muscle strength as measured by a hand-grip dynamometer. The quality of patient recovery was assessed by standardised questionnaire (Qor-40 - Quality of recovery questionnaire).

The aim was also to evaluate the applicability of the Croatian version of Qor-40 questionnaire in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ASA ( American Society of Anesthesiologists) grading status I-III
* scheduled for lumbal discectomy under general anesthesia
* signed informed consent for participating in the research

Exclusion Criteria:

* neuromuscular disease
* poorly controlled chronic or acute cardiovascular, respiratory or autoimmune disease
* allergic reaction to any of the medications in protocol
* pregnancy
* refusal to participate in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength | perioperative
  Change in muscle strength between groups measured my hand-grip dynamometer on three occasions: before general anesthesia, in the early post-anesthesia period in the operating room, and 24 hours after anesthesia.
Change in quality of patient recovery | up to 24 weeks
  Change in quality of recovery between groups measured with Qor-40 questionnaire.
  The quality of patient recovery was assessed with a Qor-40 questionnaire before anesthesia, 24 hours after anesthesia, and 30 days after anesthesia and surgery.

SECONDARY OUTCOMES:
Validation of Croatian version of the quality of recovery questionnaire (Qor-40) | perioperative
  Translate to croatian language the quality of recovery questionnaire according to Beaton and Bullinger docrtine and evaluate the applicability of the Croatian version of Qor-40 questionnaire in clinical practice in croatian speaking area

CONTACTS AND LOCATIONS:
Locations (1):
- UHCZagreb, Zagreb, Croatia

REFERENCES:
- [Result] Fuchs-Buder T, Schmartz D. [Residual neuromuscular blockade]. Anaesthesist. 2017 Jun;66(6):465-476. doi: 10.1007/s00101-017-0325-1. German. PMID 28573344
- [Result] Naguib M, Flood P, McArdle JJ, Brenner HR. Advances in neurobiology of the neuromuscular junction: implications for the anesthesiologist. Anesthesiology. 2002 Jan;96(1):202-31. doi: 10.1097/00000542-200201000-00035. No abstract available. PMID 11753022
- [Result] Srivastava A, Hunter JM. Reversal of neuromuscular block. Br J Anaesth. 2009 Jul;103(1):115-29. doi: 10.1093/bja/aep093. Epub 2009 May 24. PMID 19468024
- [Result] Jellish WS, Brody M, Sawicki K, Slogoff S. Recovery from neuromuscular blockade after either bolus and prolonged infusions of cisatracurium or rocuronium using either isoflurane or propofol-based anesthetics. Anesth Analg. 2000 Nov;91(5):1250-5. doi: 10.1097/00000539-200011000-00037. PMID 11049917
- [Result] Sweeney BP. Neuromuscular blockade and minimal monitoring. Anaesthesia. 2010 Mar;65(3):308. doi: 10.1111/j.1365-2044.2010.06252.x. No abstract available. PMID 20236270
- [Result] Gatke MR, Viby-Mogensen J, Rosenstock C, Jensen FS, Skovgaard LT. Postoperative muscle paralysis after rocuronium: less residual block when acceleromyography is used. Acta Anaesthesiol Scand. 2002 Feb;46(2):207-13. doi: 10.1034/j.1399-6576.2002.460216.x. PMID 11942873
- [Result] Desai A, Bekelis K, Ball PA, Lurie J, Mirza SK, Tosteson TD, Zhao W, Weinstein JN. Spine patient outcomes research trial: do outcomes vary across centers for surgery for lumbar disc herniation? Neurosurgery. 2012 Oct;71(4):833-42. doi: 10.1227/NEU.0b013e31826772cb. PMID 22791040
- [Result] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Result] Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, Pemberton E, Dharmage S. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003 Nov;99(5):1158-65. doi: 10.1097/00000542-200311000-00024. PMID 14576554